CLINICAL TRIAL: NCT02802891
Title: Projeto JOIN - o ar Como Meio de prevenção e a diagnóstico da Asma e Alergia
Brief Title: The JOIN Project: The Air in Diagnosis and Prevention of Asthma and Allergy
Acronym: JOIN
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Other Study IDs: SFRH/BD/108605/2015
Record Dates: First submitted 2016-06-03; First posted 2016-06-16 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-09

CONDITIONS: Asthma; Atopy
Keywords: Asthma; Allergy; Diagnosis; Endocrine disruptors; Children
MeSH Terms: conditions — Asthma; Hypersensitivity; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Exhaled breath condensate (no DNA)
  Urine (DNA)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Recruitment group: Group of individuals (aged 6 to 18 years old) recruited for the JOIN project. Consent was obtained from legal guardians for individuals under 18.
  Exclusion criteria:
  * Individuals who refused to partake in the clinical assessment, despite the legal guardians consent.
  * Individuals who provided an insufficient amount of sample (ex: low volume of EBC)

SUMMARY:
The JOIN project combines the health and indoor environment research areas to contribute in the development and validation of a new asthma diagnosis method through exhaled VOC analysis. This method is more sensitive, more specific, and completely non-invasive. Moreover, the JOIN project will assess the impact of exposure to the indoor environment, namely endocrine disruptors, on asthma and allergy development in children.

DETAILED DESCRIPTION:
Objectives:

The JOIN project combines the health and indoor environment research areas to contribute in the development and validation of a new asthma diagnosis method through exhaled VOC analysis. This method is more sensitive, more specific, and completely non-invasive. Moreover, the JOIN project will assess the impact of exposure to the indoor environment, namely endocrine disruptors, on asthma and allergy development in children. The specific objectives of the project are:

1. Classify children with asthma and healthy controls using exhaled VOC profiles;
2. Classify asthma phenotypes using exhaled VOCprofiles;
3. Evaluate the influence of prolonged exposure to exogenous VOCs on the exhaled breath samples;
4. Characterize indoor exposure by measuring the concentrations of a set of chemicals identified as EDCs in indoor air and dust at homes;
5. Evaluate the association between exposure to EDCs indoors and children's health outcomes focused on asthma/allergies and also with the exacerbation of allergies and respiratory symptoms in those who are already sensitized;
6. Investigate which building materials and consumer products might be contributing most to children's exposure;
7. Assess the association between EDCs indoor exposure and lung function, airway inflammation and responsiveness, and exhaled and urine biomarkers of disease.

The completion of this project may contribute to the validation of a new asthma diagnostic method on its way to be introduced in a real clinical context.

The indoor air quality auditing will permit a better understanding of the exposure process to endocrine disruptors and health effects, mainly in children. The project will also evaluate and compare EDCs in indoor air and in children, as a result from exposure.

Workplan:

1. Selection and recruitment of the study population

   In this project, 75 children aged 6 to 18 years old are expected to be recruited (with their legal guardian's consent) during clinical visits at the immunoallergology department of Hospital S. João. All participants will be informed about the aims and procedures of the project and will be asked to sign an informed consent form. Data collected will be confidential and participants will have the right to have their data removed from the study at any time.

   Upon agreement with the legal guardians, the visits to participants' homes will be scheduled. During the visits, EBC and urine samples will be collected, as well as exhaled breath (non-condensed).
2. Questionnaire survey A self-administered standardized questionnaire, based on International study of Asthma and Allergies in Childhood (ISAAC), completed by parents/legal guardians at home, will be carried out. Socio-demographic and economic information, smoking and drinking habits, use of personal care products, family history of diseases and dietary habits will be collected. A set of questions about respiratory/allergic health of the child, current symptoms/diagnosis (during the past 3 months) will also be included. Simultaneously, features of indoor environment factors, such as type of dwelling, age of the building, type of flooring, ventilation, will be identified.
3. Clinical assessment and biological samples collection Children attending S. João Hospital Centre for an immunoallergology clinical evaluation will be invited to participate in this study. Upon acceptance, data from spirometry, fractional exhaled nitric oxide (FeNO) and skin-prick-tests will be retrieved from the participants' clinical file. Immediately after the clinical assessment, exhaled breath condensate (EBC) will be collected from the children by breathing 10 to 15 minutes to an exhaled air condensing system (portable TurboDECCS). The EBC samples will be stored at -80ºC until laboratory analysis.

   During the indoor air quality auditing in children homes, additional EBC samples will be collected (to understand if there were significant differences when compared to the samples obtained at the hospital), as well as exhaled air (non-condensed). The exhaled air will be collected using 1 L Tedlar® bags (SKC Inc. USA) previously cleansed with 3 nitrogen flushes according to manufacturer instructions. The breathing bags serve solely to store and transport the air and are an already developed and approved product. The participants will be asked not to ingest food or flavoured beverages in the 2h prior to breath collection. Children will be instructed to cleanse their mouths with water, inhale, hold their breath for 5 seconds and subsequently exhale deeply into the Tedlar bag.

   Samples of urine will be collected from children in two moments. The 1st moment will be on the day next to clinical evaluation in S. João Hospital Centre and the 2nd moment will be on the day of indoor air quality audit.It will be previously given to each participant a commercial polypropylene specimen collection containers to obtain 6-10 mL of urine. Urine samples will be collected at home in early morning after a fasting period of at least 8 hoursto measure urinary EDCs' metabolites, such as MBzP, MEP, MEHP. After collection urine samples should be stored a -20°C and delivered on the day of indoor air quality audit. Subsequently, the samples will be frozen at -20ºC until analysis.

   Clinical diagnosis of asthma (reference standard) will be conducted by 7 different allergologists attributed randomly to each patient.
4. Building inspection and characterization A checklist will be used to get information regarding possible indoor sources (consumer and cleaning products, furniture, type of flooring), other building characteristics (e.g. age, ventilation, etc.), recent refurbishing and outdoor sources, occupant's behaviours and information on the presence of specific materials and consumers use will also be collected.
5. Indoor air audit EDCs will be measured in indoor air and dust because indoor air has been identified as an important source of chemical exposure, while house dust has been demonstrated to be an important exposure pathway. Dust also provides a record of chemicals that have been used in the home historically since degradation processes indoors are typically slow. The chemicals targeted for analysis included phthalates, bisphenol A, ethanolamines and glycol ethers. These compounds were selected based on evidence of endocrine disruption, asthma exacerbation, expected presence indoors and in consumer products, and compatibility with analytical methods developed in household exposure studies.

   EDCs indoor air samples will be collected using a URG personal pesticide sampling cartridges (University Research Glassware; chapel HilL, Nc), which will be placed in the children bedroom at approximately breathing height. At the end of the sampling period, the URG samplers will be stored at -4°c prior to shipping to the laboratory. To measure EDCs in dust, household vacuum cleaner bags will be used. Dust samples will be collected from all surfaces of the bedroom floor and also from the surface of objects, such as shelves, cupboards, doorframes, window frames, TV and audio sets, and personal computers. Dust from each bag will be sieved with a 100µm metal screen and stored in glass jars (pre-cleaned with hexane) at -20°C until chemical analysis be performed.

   Indoor air VOCs in the children bedrooms will be collected by active sampling, according to standardized procedures, at the same time as the clinical assessment in order to evaluate the influence of the pertinent ambient VOCs in the clinical test. The sampling will be performed using a 5 L flow control pump (SKC Inc. USA) connected to a stainless steel sorption tube filled with 200 mg of Tenax TA 60/80 (Supelco). The sampling will start at the same time as the clinical assessment and will be programmed to end after one hour, giving a representative sample of the indoor air VOCs at the time of the exhaled breath collection. At the end of the sampling, the tubes will be sealed with air-tight caps and transported to the laboratory, where they will be stored at room temperature until analysis.
6. Laboratory analysis Volatile organic compounds and EDCs will be analysed by electronic nose (Cyranose 320). Multivariate analysis will be performed to observe if VOC profiles of participants with asthma is different from those without asthma. Classification rates, area under the ROC curve, sensitivity and specificity will be estimated for the different models.

ELIGIBILITY:
Inclusion Criteria:

* Individuals (6 to 18 years old) with skin prick tests and spirometry with bronchodilation results.

Exclusion Criteria:

* Individuals with chronic diseases (other than asthma and atopy)
* Planning to change home address in the next 4 months
* Low volume of EBC
* Refused to participate despite signing written consent

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children performing skin prick tests and spirometry with bronchodilation while attending immunoallergology consultations in the outpatients clinic of S. João Hospital Centre.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-09-13 (Actual); Study Completion 2017-09-13 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds in the exhaled breath condensate | 4 to 8 months after recruitment
  Volatile organic compounds, released from EBC through heating, will be measured by an electronic nose system

SECONDARY OUTCOMES:
Endocrine disruptors in the urine | 4 to 8 months after recruitment
ISAAC-based questionnaire | 4 to 8 months after recruitment
24h food questionnaire | 4 to 8 months after recruitment
Endocrine disruptors in the house dust | 4 to 8 months after recruitment

OTHER OUTCOMES:
Skin prick tests | During recruitment
  Performed during the regular examination in the outpatient clinic. Requested by the physician.
Spirometry with bronchodilation | During recruitment
  Performed during the regular examination in the outpatient clinic. Requested by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: André Moreira, MD PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Centro Hospitalar S. João, Porto, Portugal